CLINICAL TRIAL: NCT05313347
Title: A Pilot Study to Investigate Neural Processing During Sensory Specific Satiety Using Gustatory Stimulation
Brief Title: Neural Correlates of Sensory Specific Satiety
Acronym: Gusto
Status: Completed | Type: Observational
Sponsor: University of Heidelberg Medical Center (Other)
Responsible Party: Principal Investigator, Joe Simon, Principal Investigator, University of Heidelberg Medical Center
Other Study IDs: S-656/2019-2
Record Dates: First submitted 2022-03-28; First posted 2022-04-06 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Satiety Response; Functional Neuroimaging; Obesity
Keywords: fmri; sensory specific satiety
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healty Participants with varying BMI: 30 healthy participants with a body mass index ranging from 17.5 to 35kg/m2.

SUMMARY:
Sensory specific satiety, or the phenomenon that the pleasantness of a particular taste declines when certain types food are consumed to satiety, plays an important role in food choice and meal termination.The rewarding effect of sugar will be investigated in a group of 30 healthy participants with a body mass index ranging from 17.5 to 35kg/m2. A gustatory stimulation paradigm designed to induce sensory specific satiety for glucose will be employed. The aim is to assess neuronal stimulus processing in relation to the sensory satiety level and to investigate the relationship with everyday eating behavior.

DETAILED DESCRIPTION:
Sensory specific satiety, or the phenomenon that the pleasantness of a particular taste declines when certain types food are consumed to satiety, plays an important role in food choice and meal termination. Since changes in taste, smell and appetite are commonly observed in obesity, previous studies investigated the relation of sensory specific satiety to weight gain, but observed conflicting results. To gain a more detailed understanding of the relationship between sensory specific satiety and weight homeostasis, we will examine the rewarding effect of sugar in a group of 30 healthy participants with a body mass index ranging from 17.5 to 35kg/m2. We will employ a gustatory stimulation paradigm designed to induce sensory specific satiety for glucose. During fMRI scanning, glucose and water are applied orally using a gustometer. Furthermore, relevant hormonal satiety parameters are measured, as well as dietary behavior and food preferences in everyday life. This will allow us to assess neuronal stimulus processing in relation to the sensory satiety level and to investigate the relationship with everyday eating behavior. A better understanding of factors contributing to the development and maintenance of overweight are crucial for the development of new treatment options for obesity.

ELIGIBILITY:
Inclusion Criteria:

1. BMI between 17,5 and 35 kg/m².
2. Over age of 18 years.
3. Right-handedness.
4. Normal or corrected-to-normal vision.
5. Capacity to consent.

Exclusion Criteria:

1. History of head injury or surgery.
2. History of neurological disorder.
3. Severe psychiatric comorbidity.
4. Lifetime or current medical illness that could potentially affect appetite or weight (including eating disorders diagnosis)
5. Smoking.
6. Current psychotropic medication.
7. Inability to undergo fMRI scan (e.g. metallic implants, claustrophobia, pacemakers).
8. Pregnancy.

Ages: 18 Years to 55 Years | Sex: All
Age Groups: Adult
Study Population: Healthy controls with BMI between 17,5 and 35 kg/m².
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-10-01 (Actual)

PRIMARY OUTCOMES:
Choice of water compared to choice of sugar during Sensory Specific Satiety. | 1 hour
  Comparing tasting of water with tasting of sugar (G10%) when participants are allowed to freely chose between the two during specific satiety for sugar.
Choice of water compared to passive ingestion of 20% sugar solution during Sensory Specific Satiety. | 1 hour
  Comparison of voluntary tasting of water with the "forced" tasting of sugar during specific satiety for sugar.

SECONDARY OUTCOMES:
Influence of variations in BMI on brain activation during Sensory Specific Satiety. | 1 hour

CONTACTS AND LOCATIONS:
Overall Officials: joe simon, Ph.D., Principal Investigator — Heidelberg University
Locations (1):
- University Hospital Heidelberg, Heidelberg, Germany

IPD SHARING:
Plan to Share IPD: No